CLINICAL TRIAL: NCT04142619
Title: Phase I, Open-label Dose-escalation Study to Evaluate the Safety, Expansion, Persistence and Clinical Activity of UCARTCS1A (Allogenic Engineered T-cells Expressing Anti-CS1 Chimeric Antigen Receptor) Administered in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study Evaluating Safety and Efficacy of UCART Targeting CS1 in Patients With Relapsed/Refractory Multiple Myeloma (MELANI-01)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was discontinued due to sponsor's decision and not a consequence of any safety concern.
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCARTCS1A_01
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Chimeric Antigen Receptor T-Cell (CART-T) therapy; Transcription Activator-Like Effector Nuclease (TALEN); Allogeneic
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Several tested doses of UCARTCS1A until the Maximum Tolerated Dose (MTD) is identified.
  Interventions: Biological: UCARTCS1A

INTERVENTIONS:
Biological: UCARTCS1A — Allogenic engineered T-cells expressing anti- CS1 Chimeric Antigen Receptor

SUMMARY:
This is a Phase I, FIH, open-label, dose escalation study evaluating Safety and Efficacy of UCART targeting CS1 in patients with Relapsed or Refractory Multiple Myeloma (MM). The purpose of this study is to evaluate the safety and clinical activity of UCARTCS1A and to determine the Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of active multiple myeloma (as defined by International Myeloma Working Group [IMWG] criteria) who have relapsed/refractory disease after and have received at least 3 prior lines of prior therapy.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1;
* No previous treatment with investigational gene targeting CS1 or chimeric antigen receptor therapy targeting CS1
* Adequate organ function, including bone marrow, renal, hepatic, pulmonary, and cardiac function based on the last assessment performed within the screening period.
* Other criteria may apply.

Exclusion Criteria:

* Previous treatment with investigational gene therapy targeting CS1 or chimeric antigen receptor therapy targeting CS1;
* Any cellular therapy (other than autologous or allogenic HSCT) within 60 days prior to enrollment;
* Prior treatment with rituximab or other anti-CD20 therapy within 3 months
* Any known active or uncontrolled infection
* Autologous hematopoietic stem cell transplantation (HSCT) within 12 weeks prior to enrollment; any cellular therapy (other than autologous) within 60 days prior to enrollment; prior allogeneic HSCT.
* Seropositive for Hepatitis C virus or positive for Hepatitis B surface antigen or core antibody.
* Presence of active and clinically relevant central nervous system disorder, such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, or organic brain syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Safety of UCARTCS1A | 24 months.
  Incidence, nature and severity of adverse events and serious adverse events (SAEs) throughout the study.

SECONDARY OUTCOMES:
Response Assessment | 24 months
  At Day 35, Day 56 (M2), Day 84 (M3), Follow-up [Q3M up to Month 24; i.e., Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21 and Month 24
Duration of Response | 24 months
  Time Frame: From the date of the initial response to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24]
Progression Free Survival | 24 months
  From the first day of study treatment to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24
Overall Survival | 24 months
  From the first day of study treatment to the date of death from any cause, assessed up to Month 24

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSF Medical Center- Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sarah Cannon Research Institute - Colorado Blood Cancer Institute, Denver, Colorado
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Mayo Clinical Cancer Center (MCCC), Rochester, Minnesota
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Sarah Cannon Research Institute - Methodist Healthcare, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No